CLINICAL TRIAL: NCT00200967
Title: Asthma Clinical Research Network (ACRN) Trial - Long-Acting Beta Agonist Response by Genotype (LARGE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Asthma Clinical Research Network (Network)
Responsible Party: Principal Investigator, Vernon M. Chinchilli, PhD, Professor and Chair, Department of Public Health Sciences, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 262; 5U10HL074231 (NIH); U10HL074073 (NIH); U10HL074204 (NIH); U10HL074208 (NIH); U10HL074212 (NIH); U10HL074218 (NIH); U10HL074225 (NIH); U10HL074227 (NIH); U10HL074231 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Salmeterol Xinafoate; Beclomethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B16 Arg/Arg (Experimental): B16 Arg/Arg genotype Sequence 1: inhaled salmeterol + inhaled beclomethasone hydroflouroalkane (HFA), followed by inhaled placebo salmeterol + inhaled beclomethasone HFA Sequence 2: inhaled placebo salmeterol + inhaled beclomethasone HFA, followed by inhaled salmeterol + inhaled beclomethasone HFA
  Interventions: Drug: salmeterol; Drug: beclomethasone HFA
- B16 Gly/Gly (Experimental): B16 Gly/Gly genotype Sequence 1: inhaled salmeterol + inhaled beclomethasone HFA, followed by inhaled placebo salmeterol + inhaled beclomethasone HFA Sequence 2: inhaled placebo salmeterol + inhaled beclomethasone HFA, followed by inhaled salmeterol + inhaled beclomethasone HFA
  Interventions: Drug: salmeterol; Drug: beclomethasone HFA

INTERVENTIONS:
Drug: salmeterol — 50 micrograms (mcg) twice per day (BID) (Serevent 50 mcg diskus, GlaxoSmithKline (GSK), North Carolina)
  Other Names: Serevent
Drug: beclomethasone HFA — 240 mcg beclomethasone HFA (QVAR, Teva Pharmaceutical Industries)
  Other Names: QVAR

SUMMARY:
The purpose of this trial is to determine whether regularly scheduled use of an inhaled long-acting beta agonist (salmeterol) in the setting of concomitant use of inhaled corticosteroids (beclomethasone hydroflouroalkane (HFA) inhaler) will have a detrimental effect on asthma control in people who bear the B16-Arg/Arg genotype of the beta-2 adrenergic receptor gene, as compared to people with asthma of similar severity who bear the B16-Gly/Gly genotype.

DETAILED DESCRIPTION:
BACKGROUND:

The purpose of this study is to compare the effects of a long-acting beta agonist in patients with asthma receiving inhaled corticosteroids who express two distinct polymorphisms of the beta-2 adrenergic receptor.

DESIGN NARRATIVE:

Participants were homozygous for arginine or glycine at the 16th amino-acid position of the β-2 adrenergic receptor (B16 Arg/Arg or B16 Gly/Gly). Individuals were matched against their opposite genotype by forced expiratory volume in one second (FEV1) and race. Matched participants entered an 8-week run-in period. This is a 62-week crossover design where subjects receive the following therapies:

* Beclomethasone HFA (240 µg twice a day (BID)) + as-needed (PRN) albuterol: 8-week run-in
* Beclomethasone HFA (240 µg BID) + salmeterol (50 µg BID) + PRN ipratropium bromide + PRN albuterol: 18-week treatment period
* Beclomethasone HFA (240 µg BID) + PRN albuterol: 8-week run-out
* Beclomethasone HFA (240 µg BID) + placebo salmeterol + PRN ipratropium bromide + PRN albuterol: 18-week treatment period
* Beclomethasone HFA (240 µg BID) + PRN albuterol: 10-week run-out

The order of treatments received during the two treatment periods is randomized.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 18 and older
* Clinical history consistent with asthma
* For subjects regularly using inhaled corticosteroids, FEV1 50% of predicted, methacholine PC20 FEV1 16 mg/ml or 12% and 200 ml, improvement in FEV1 after 2 puffs of inhaled albuterol
* For subjects not regularly using inhaled corticosteroids, FEV1 40% of predicted, methacholine PC20 FEV1 8 mg/ml or 12% and 200 ml, improvement in FEV1 after 2 puffs of inhaled albuterol
* Genotype eligibility (determined during screening)

Exclusion Criteria:

* Smoker (total smoking history must be less than 10 pack years)
* Significant unstable medical condition other than asthma
* History of life-threatening asthma requiring treatment with intubation and mechanical ventilation in the past 10 years
* Pregnant or lactating

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2004-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Homer Boushey, Principal Investigator — University of California, San Francisco; Mario Castro, Principal Investigator — Washington University School of Medicine; Vernon M. Chinchilli, PhD, Principal Investigator — Milton S. Hershey Medical Center; Elliot Israel, Principal Investigator — Brigham and Women's Hospital; Robert Lemanske, Principal Investigator — University of Wisconsin, Madison; Richard Martin, Principal Investigator — National Jewish Medical & Research Center; Stephen Peters, Principal Investigator — Wake Forest University Health Sciences; Stephen Wasserman, Principal Investigator — University of California, San Diego
Locations (7):
- United States (7):
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - National Jewish Medical & Research Center, Denver, Colorado
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Washington University, St Louis, Missouri
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Wisconsin Madison, Madison, Wisconsin

REFERENCES:
- [Result] Wechsler ME, Kunselman SJ, Chinchilli VM, Bleecker E, Boushey HA, Calhoun WJ, Ameredes BT, Castro M, Craig TJ, Denlinger L, Fahy JV, Jarjour N, Kazani S, Kim S, Kraft M, Lazarus SC, Lemanske RF Jr, Markezich A, Martin RJ, Permaul P, Peters SP, Ramsdell J, Sorkness CA, Sutherland ER, Szefler SJ, Walter MJ, Wasserman SI, Israel E; National Heart, Lung and Blood Institute's Asthma Clinical Research Network. Effect of beta2-adrenergic receptor polymorphism on response to longacting beta2 agonist in asthma (LARGE trial): a genotype-stratified, randomised, placebo-controlled, crossover trial. Lancet. 2009 Nov 21;374(9703):1754-64. doi: 10.1016/S0140-6736(09)61492-6. PMID 19932356
- See also: Asthma Clinical Research Network (ACRN) Website — http://www.acrn.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the LARGE trial began in November 2004 and the final participant visits occurred in February 2008. Seven academic medical centers throughout the US recruited the participants.
Pre-assignment Details: 474 participants were screened: 78 had B16 Arg/Arg genotype; 166 had B16 Gly/Gly genotype; 230 had Arg/Gly genotype. 47 matched Arg/Arg-Gly/Gly pairs entered the 8-week run-in period. 42 Arg/Arg were randomized (2 withdrew, 2 noncompliant, 1 lost); 45 Gly/Gly were randomized (1 withdrew, 1 noncompliant).
Groups:
- B16 Arg/Arg; B16 Gly/Gly: B16 Arg/Arg genotype Sequence 1: inhaled salmeterol + inhaled beclomethasone HFA, followed by inhaled placebo salmeterol + inhaled beclomethasone HFA Sequence 2: inhaled placebo salmeterol + inhaled beclomethasone HFA, followed by inhaled salmeterol + inhaled beclomethasone HFA
Period: First Treatment Period
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Started | 42 | 45
First Treatment Period | 42 | 45
Completed | 36 | 44
Not Completed | 6 | 1
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Pregnancy | 1 | 0
Period: Wash-out Period
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Started | 36 | 44
Completed | 36 | 43
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: Second Treatment Period
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Started | 36 | 43
Completed | 35 | 41
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Run-out Period
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Started | 35 | 41
Completed | 34 | 41
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | B16 Arg/Arg | B16 Gly/Gly | Total
Number analyzed (Participants) | 42 | 45 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 42 | 45 | 87
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (11) | 42 (12) | 41 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 10 | 16 | 26
Region of Enrollment [Number; unit: participants]
  United States | 42 | 45 | 87.0

OUTCOME MEASURES:

1. Primary Outcome: Morning (AM) Peak Expiratory Flow (PEF) Rate
Description: Change between placebo salmeterol and active salmeterol for AM PEF rate
Time Frame: Measured daily using a hand-held peak flow meter, and then averaged between weeks 0, 2, 6, 10, 14, and 18 of each treatment period
Population: An intention-to-treat (ITT) paradigm was invoked in which the available data (without any imputation for missing data) on all randomized participants were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: liters per minute
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
liters per minute | -21 [-31 to -12] | -22 [-32 to -11]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; A mixed-effects linear model was applied to account for the repeated measurements within each treatment period of the crossover design. A sample size of 40 participants per genotype was required to detect a difference of 25 L/min in AM PEF (and relevant effect sizes for secondary outcomes) with a two-sided, 0.05 significance level test with 90% statistical power and a 15% drop-out rate; Test type: Superiority or Other; p = 0.99, Mixed Models Analysis; Mean Difference (Final Values) = 0, 95% CI [-14 to 14], Standard Error of Mean 7 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for AM PEF rate

2. Secondary Outcome: Evening (PM) Peak Expiratory Flow (PEF) Rate
Description: Change between placebo salmeterol and active salmeterol for PM PEF rate
Time Frame: as for outcome 1
Population: An ITT paradigm was invoked in which the available data (without any imputation for missing data) on all randomized participants were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: liters per minute
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
liters per minute | -25 [-34 to -16] | -24 [-34 to -14]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; A mixed-effects linear model was applied to account for the repeated measurements within each treatment period of the crossover design; Test type: Superiority or Other; p = 0.82, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI [-15 to 12], Standard Error of Mean 7 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for PM PEF rate

3. Secondary Outcome: Peak Expiratory Flow (PEF) Variability
Description: Change between placebo salmeterol and active salmeterol for PEF variability, where PEF variability is defined as 100% x (PM PEF - AM PEF)/(PM PEF)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
percentage | 0.2 [-0.6 to 1.0] | 0.7 [0.0 to 1.4]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.31, Mixed Models Analysis; Mean Difference (Final Values) = -0.6, 95% CI [-1.6 to 0.5], Standard Error of Mean 0.5 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for PEF variability

4. Secondary Outcome: Asthma Symptoms
Description: Change between placebo salmeterol and active salmeterol for asthma symptoms (0=absent, 1=mild, 2=moderate, 3=severe).
Time Frame: Recorded daily on a diary card, and then averaged between weeks 0, 2, 6, 10, 14, and 18 of each treatment period
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
units on a scale | 0.04 [0.00 to 0.12] | 0.00 [-0.01 to 0.02]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; A mixed-effects linear model was attempted but could not converge because very few symptoms were recorded, so a nonparametric analysis was applied; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.02, 95% CI [-0.02 to 0.07], Standard Error of Mean 0.02 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for asthma symptoms

5. Secondary Outcome: Rescue Medication (Ipratropium and Albuterol) Use
Description: Change between placebo salmeterol and active salmeterol for rescue medication use
Time Frame: Recorded daily on a diary card, and then averaged between weeks 0, 2, 6, 10, 14, and 18 of each treatment period
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: puffs per day
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
puffs per day | 0.2 [0.0 to 0.5] | 0.0 [0.0 to 0.2]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; A mixed-effects linear model was attempted but could not converge because very few usages of rescue medications were recorded, so a nonparametric analysis was applied; Test type: Superiority or Other; p = 0.25, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.0, 95% CI [-0.1 to 0.2], Standard Error of Mean 0.1 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for rescue medication use

6. Secondary Outcome: Spirometry Forced Expiratory Volume in One Second (FEV1), Pre-bronchodilator
Description: Change between placebo salmeterol and active salmeterol for Spirometry FEV1, pre-bronchodilator
Time Frame: Clinic visits at weeks 0, 2, 6, 10, 14, and 18 of each treatment period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
liters | -0.08 [-0.13 to -0.03] | -0.04 [-0.09 to 0.00]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.34, Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI [-0.10 to 0.03], Standard Error of Mean 0.03 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for Spirometry FEV1, pre-bronchodilator

7. Secondary Outcome: Spirometry Forced Vital Capacity (FVC), Pre-bronchodilator
Description: Change between placebo salmeterol and active salmeterol for Spirometry FVC, pre-bronchodilator
Time Frame: Clinic visits at weeks 0, 2, 6, 10, 14, and 18 of each treatment period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
liters | -0.04 [-0.08 to 0.01] | -0.03 [-0.09 to 0.03]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.91, Mixed Models Analysis; Mean Difference (Final Values) = 0.00, 95% CI [-0.08 to 0.07], Standard Error of Mean 0.03 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for Spirometry FVC, pre-bronchodilator

8. Secondary Outcome: Spirometry Peak Expiratory Flow (PEF) Rate, Pre-bronchodilator
Description: Change between placebo salmeterol and active salmeterol for Spirometry PEF rate, pre-bronchodilator
Time Frame: Clinic visits at weeks 0, 2, 6, 10, 14, and 18 of each treatment period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: liters per minute
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
liters per minute | -17 [-27 to -8] | -17 [-27 to -6]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.93, Mixed Models Analysis; Mean Difference (Final Values) = -1, 95% CI [-15 to 14], Standard Error of Mean 7 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for Spirometry PEF rate, pre-bronchodilator

9. Secondary Outcome: Exhaled Nitric Oxide (eNO)
Description: Change between placebo salmeterol and active salmeterol for eNO
Time Frame: Clinic visits at weeks 0, 2, 6, 10, 14, and 18 of each treatment period
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: parts per billion
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
parts per billion | 0.12 [-0.01 to 0.24] | -0.02 [-0.15 to 0.11]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; A mixed-effects linear model was applied to the natural logarithm of eNO to account for the repeated measurements within each treatment period of the crossover design; Test type: Superiority or Other; p = 0.13, Mixed Models Analysis; Mean Difference (Final Values) = 0.14, 95% CI [-0.04 to 0.31], Standard Error of Mean 0.08 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for eNO

10. Secondary Outcome: Exhaled Breath Condensate (EBC)
Description: Change between placebo salmeterol and active salmeterol for EBC
Time Frame: Clinic visits at weeks 0, 10, and 18 of each treatment period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: pH
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
pH | -0.10 [-0.45 to 0.26] | -0.03 [-0.37 to 0.31]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.79, Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 95% CI [-0.56 to 0.43], Standard Error of Mean 0.24 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for EBC

11. Secondary Outcome: Methacholine Provocative Concentration 20 (PC20)
Description: Change between placebo salmeterol and active salmeterol for methacholine PC20
Time Frame: Clinic visits at weeks 0 and 18 of each treatment period
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: milligrams per milliliter
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
milligrams per milliliter | 0.06 [-0.60 to 0.71] | -1.27 [-1.87 to -0.66]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; A mixed-effects linear model was applied to the base-2 logarithm of the methacholine PC20 to account for the repeated measurements within each treatment period of the crossover design; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Final Values) = 1.32, 95% CI [0.43 to 2.21], Standard Error of Mean 0.45 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for methacholine PC20

12. Secondary Outcome: Asthma Control Questionnaire (ACQ)
Description: Change between placebo salmeterol and active salmeterol for ACQ, where ACQ ranges from 0 (best asthma control) to 6 (worst asthma control).
Time Frame: Clinic visits at weeks 0 and 18 of each treatment period
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Number analyzed (Participants) | 42 | 45
units on a scale | 0.13 [-0.06 to 0.32] | 0.11 [-0.04 to 0.26]
Statistical Analysis 1: Comparison: B16 Arg/Arg vs B16 Gly/Gly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.89, Mixed Models Analysis; Mean Difference (Final Values) = 0.02, 95% CI [-0.23 to 0.26], Standard Error of Mean 0.12 — The comparison represents the difference between Arg/Arg and Gly/Gly participants based on the change between placebo salmeterol and active salmeterol for ACQ

ADVERSE EVENTS:
Time Frame: 1 year
Description: does not differ from clinicaltrials.gov definitions
Arm/Group | B16 Arg/Arg | B16 Gly/Gly
Serious Adverse Events (participants affected / at risk) | 1/42 | 4/45
Other Adverse Events (participants affected / at risk) | 20/42 | 20/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B16 Arg/Arg (N=42) | B16 Gly/Gly (N=45)
hospitalization (General disorders) | 0 (0) | 1 (1)
hospitalization (Psychiatric disorders) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B16 Arg/Arg (N=42) | B16 Gly/Gly (N=45)
respiratory infection (Respiratory, thoracic and mediastinal disorders) | 20 (100) | 20 (98)

LIMITATIONS AND CAVEATS:
The study used a moderately high dose of ICS. Genotype-specific effects may be evident at lower doses of ICS often used in combination therapy. Also, short-acting β2-agonists have been shown to have genotype-specific effects on asthma outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No